CLINICAL TRIAL: NCT00001110
Title: Effect of Highly Active Antiretroviral Therapy (HAART) on Viral Burden and Immune Function in the Lungs of HIV-Infected Subjects
Brief Title: Effect of Anti-HIV Therapy (HAART) on HIV Levels in the Lungs and on Lung Cell Inflammation in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 723; AACTG 723; 10188 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: Lung; HIV-1; Viremia; Anti-HIV Agents; Viral Load; Bronchoalveolar Lavage Fluid
MeSH Terms: conditions — HIV Infections; Viremia | interventions — Bronchoalveolar Lavage

INTERVENTIONS:
Procedure: Bronchoalveolar lavage

SUMMARY:
The purpose of this study is to see: (1) how the amount of HIV in the lungs compares to that in the blood; (2) if HAART reduces the amount of HIV in the lungs; and (3) if HAART reduces lung inflammation in HIV-infected patients.

Lung-cell inflammation in HIV-infected patients is probably caused by HIV infection of these cells. The amount of inflammation may correspond to the amount of HIV (viral load) in the lungs (i.e., mild inflammation indicates a low amount of HIV; severe inflammation indicates a high amount of HIV). HAART is used to decrease the amount of HIV in the body. If HAART is able to decrease viral load in the lungs, it should also be able to decrease lung-cell inflammation in these patients.

DETAILED DESCRIPTION:
Lymphocytic alveolitis in HIV-infected patients probably represents a local immune response to HIV-infected cells in the lung. The intensity of lymphocytic alveolitis may therefore reflect the viral load in the lung. If so, treatment that reduces viral load in the lung (e.g., HAART) should also decrease the number of cytotoxic T lymphocytes (CTLs) in the alveolar space and should return pulmonary immune responses toward normal.

Patients are stratified by CD4 count: less than 200 cells/mm3 or 200 - 500 cells/mm3. BAL is performed and blood samples are collected prior to initiation of HAART and after 1 and 6 months of HAART. If a patient has detectable HIV in the lung after 6 months of HAART, the patient is asked to submit to an optional fourth BAL after 12 months of HAART. BAL fluid and cells are analyzed for HIV viral load, percent lymphocytes, and lymphocyte subsets. Responses in the lung are compared to simultaneous changes in these variables found in the peripheral blood. Each patient serves as his/her own control.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are at least 18 years old.
* Have a CD4 count less than or equal to 500 cells/mm3 and an HIV RNA level greater than or equal to 5000 copies/ml.
* Are about to start a regimen of at least 3 anti-HIV drugs (HAART).

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have ever received protease inhibitors (PIs) or nonnucleoside reverse transcriptase inhibitors (NNRTIs).
* Have had signs or symptoms of lung disease in the past 30 days (pneumonia, bronchitis, emphysema, asthma, severe cough, or severe shortness of breath).
* Have received certain medications, including HIV vaccines.
* Have received chemotherapy within 30 days prior to study entry, or have cancer that will require chemotherapy.
* Are pregnant and will be beyond the first 3 months of pregnancy by Week 24 (Month 6) of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 1999-08; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HL Twigg, Study Chair; J Wheat, Study Chair
Locations (5):
- United States (4):
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
- Puerto Rico-AIDS CRS, San Juan, Puerto Rico